CLINICAL TRIAL: NCT05154604
Title: A Phase 1 Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-A1921 in Subjects With Advanced Malignant Solid Tumour .
Brief Title: A Study of SHR-A1921 for Injection in Subjects With Advanced Solid Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1921-I-101
Record Dates: First submitted 2021-11-12; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Advanced Solid Tumours

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group: SHR-A1921 (Experimental)
  Interventions: Drug: SHR-A1921

INTERVENTIONS:
Drug: SHR-A1921 — Treatment group: Subjects will receive an intravenous infusion of SHR-A1921 in a dose escalation until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the study.

SUMMARY:
To assess the safety and tolerability of SHR-A1921 in patients with advanced solid tumours, to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and/or recommended phase II dose (RP2D) of SHR-A1921

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent；
2. Aged 18-75 years (inclusive), males and females;
3. Consents to provide tumor tissue samples;
4. Subjects must have histologically or clinically confirmed advanced and/or metastatic malignancies for which failure of standard treatment or lack of effective standard treatment;
5. At least one measurable lesion according to RECIST v1.1;
6. ECOG score of 0-1;
7. Expected survival ≥ 12 weeks;
8. Adequate bone marrow reserve and organ function ；
9. For female patients of childbearing potential or male patients with partners of childbearing potential who are not sterilized by surgical operations, they are required to use a medically approved contraceptive measure during the study treatment period and within 3 months after the end of the study treatment; For female patients of childbearing potential who are not sterilized by surgical operations, they must have a negative serum HCG test result within 72 h prior to study enrollment; and they must not be in the lactation period;

Exclusion Criteria:

1. Known and untreated central nervous system (CNS) or leptomeningeal metastases;
2. Macrovascular invasion based on imaging;
3. Cancerous ascites, pleural effusion or pericardial effusion with clinical symptoms;
4. Has a history of a second malignancy;
5. History of immunodeficiency disease or organ transplant;
6. Uncontrolled cardiac diseases or symptoms;
7. Has a history of non-infectious ILD/pneumonitis that required steroids, or has current ILD/pneumonitis;
8. Has a history of active chronic enteritis 6 weeks prior to the initiation of the study treatment or intestinal obstruction, gastrointestinal perforation 3 months prior to the initiation of the study treatment;
9. Has a history of Grade≥2 bleeding 4 weeks prior to the initiation of the study treatment or is current receiving anticoagulation therapy;
10. Subjects with active hepatitis B or active hepatitis C;
11. Subjects who have received systemic anti-tumor treatments 4 weeks prior to the initiation of the study treatment.
12. Has unresolved toxicities from previous anticancer therapy.
13. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients of SHR-A1921;
14. Subjects with other potential factors that may affect the study results or result in the premature discontinuation as determined by the investigator, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, or family or social factors that could affect the safety of the patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | 21 Days (first cycle)
Maximum Tolerable Dose (MTD) | 21 Days (first cycle)
Recommended phase II dose (RP2D) | Screening up to dose escalation and expansion study completion, appropriately to 1 year
Adverse Events | Screening up to study completion, an average of 1 year
  Incidence and grade of adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Time to reach maximum concentration (Tmax) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Maximum concentration (Cmax) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Area under the concentration-time curve from time zero to the time of the last quantifiable time point t (AUC0-t) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-t) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Terminal half-life (t1/2) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Total body clearance (CL) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Volume of distribution at steady state (Vss) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Mean residence time (MRT) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Maximum steady-state drug concentration during a dosage interval (Css, max) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Minimum steady-state drug concentration during a dosage interval (Css, min) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Accumulation ratio (Rac) of SHR-A1921、total antibody | Screening up to end of treatment, an average of 1 year
Anti-drug antibody(ADA) level of SHR-A1921 | Screening up to 90 days after the last dose, an average of 1 year
Objective Response Rate (ORR) assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Duration of Response (DoR) assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Disease Control Rate (DCR) assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Progression-Free Survival (PFS) assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Overall Survival (OS) | Screening up to study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided